CLINICAL TRIAL: NCT01969305
Title: A Computerized Family-Based Youth HIV and Drug Abuse Prevention in Kazakhstan
Brief Title: Youth Drug Abuse Prevention in Kazakhstan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB13-0841; R34DA033201 (NIH)
Record Dates: First submitted 2013-07-06; First posted 2013-10-25 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2018-09

CONDITIONS: Drug Use
Keywords: Kazakhstan; Central Asia; HIV prevention; Adolescents; Sexual risk behaviors; Drug abuse prevention; Multi-media intervention; Drug use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kazakhstani Family Together (KFT) (Experimental): Usual Care Plus KFT: Family-based multi-media HIV and drug abuse prevention intervention
  Interventions: Behavioral: Kazakhstani Family Together
- Health education curriculum (Experimental): Usual Care Alone: Health education curriculum on HIV and drug use prevention
  Interventions: Behavioral: Usual Care Alone

INTERVENTIONS:
Behavioral: Kazakhstani Family Together — Adolescent-caregiver pairs will receive three 45-minute interactive multi-media sessions with avatars customized to participants' gender that will focus on risk reduction self-efficacy, resistance to peer pressure, decision-making skills and caregiver-adolescent communication, support and monitoring to strengthen youth's relationships with caregivers and reduce youth's risks of drug use and sexual risk behaviors. Through the multimedia tool, participants will confront a series of sexual risks and substance use related situations and will practice their listening, empathy, assertiveness, refusal, and other interpersonal skills. Each caregiver-youth pair will work jointly and engage in discussions, exercises, and behavioral rehearsal as directed by the program.
  Arms: Kazakhstani Family Together (KFT)
Behavioral: Usual Care Alone — Adolescents from both study arms will receive the usual care, a health education program about how to prevent drug use and HIV/STIs (sexually transmitted infections). The health education curriculum is delivered in a group format by trained peer educators and outreach workers. The curriculum consists of three 45-minute sessions that include lectures and interactive quizzes about drugs and HIV. These three sessions include information on the following topics:
  1. Facts and Myth about HIV. HIV/STIs modes of transmission;
  2. Prevention of HIV. Abstinence and Safe Sex. Attitudes and values about sexuality, sexual risk behaviors, and condom use;
  3. Knowledge, attitudes and beliefs about drinking and drug use. Risks and consequences of drug use.
  Arms: Health education curriculum

SUMMARY:
This pilot study will adapt and test the feasibility and estimate the effect size parameters of Kazakhstani Family Together (KFT), a family-based multi-media intervention designed to reduce sexual and drug-related risks for HIV infection among at-risk 14-17 year old females and males living in communities highly affected by heroin trade and use in Almaty, Kazakhstan.

DETAILED DESCRIPTION:
The purpose of this study is to adapt an evidence-based HIV and substance use prevention intervention for most at-risk adolescents and their caregivers (parents or other adult family members) from drug-risk communities in Kazakhstan. Located on major drug trafficking routes (between Afghanistan, the world's largest opium producer, and Russia), Central Asia and Kazakhstan, in particular, face one of the fastest growing rates of HIV infection in the world disproportionately affecting young people ages 15-29. Youth exposed to drugs at home and in the community are particularly at risk.

The country's HIV prevention efforts for youth are limited to a knowledge-based approach, which does not equip at-risk youth with skills required to deal with situations of risk exposure. Parents or other caregivers, who represent a significant protective force in a family-oriented culture of Central Asia, are largely excluded from youth prevention efforts in Kazakhstan.

KFT is a family-based multi-media intervention designed to reduce sexual and drug-related risks for HIV infection among at-risk adolescents. To address the dual risk of HIV and substance use, the proposed intervention combines empirically tested skills-based and family involvement approaches and utilizes multi-media computer technology to develop an engaging and potentially cost-effective tool with high fidelity and easy scalability. During each of the sessions, youth and caregivers will participate in interactive computer activities to learn skills and have conversations focused on risky behaviors.

During the development stage, the US and Kazakhstani investigative team will conduct formative research and will work closely with the local Community Collaborative Board to adapt the intervention to the cultural context of at-risk families in Kazakhstan.

Further, the KFT intervention will be tested in a pilot Randomized Controlled Trial with 248 adolescents and 248 of their caregivers. Intervention arm adolescent-caregiver pairs will receive three 45-minute interactive multi-media sessions with avatars customized to participants' gender that will focus on risk reduction self-efficacy, resistance to peer pressure, and caregiver-adolescent communication, support and monitoring. Adolescents from both intervention and control arms will receive the usual care services available for at-risk youth, which includes health education sessions on HIV and drug use delivered by peer educators and outreach workers.

ELIGIBILITY:
Inclusion Criteria:

1. Youth are between the ages of 14-17.
2. Youth exhibits one of the following risk factors: substance-using peers or friends, parental history of drug use, parental history of alcohol problems, parental criminal history, adolescent's history of drug use, running away from home, school drop-out or history of sexual activity.
3. You and caregiver are able to speak and read Russian.
4. Both youth and caregiver (parent or other caregiving adult family member) can commit to study participation.
5. Youth and caregiver do not plan to move in the next 6 months.

Exclusion Criteria:

1. Youth are under the age of 14 or over the age of 17.
2. Youth does not exhibit one of the aforementioned risk factors.
3. Youth and caregiver do not speak and read Russian.
4. Youth and caregiver are unable to commit to study participation.
5. Youth or caregiver has plans to move within the next 6 months.
6. Youth or caregiver has a cognitive impairment.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in onset and 30-day alcohol and drug use from baseline to 6 months | Up to 6-months
  Measures will ask youth to report the frequency and quantity of alcohol and drug use in the past 30 days (number of alcoholic drinks, puffs of marijuana, or initiation of injection drug use). Substance use includes specific probes, including street names for alcohol, marijuana, ecstasy, cocaine, injecting drug use, heroin, inhalants, hallucinogens, and other drugs as appropriate to the context.

SECONDARY OUTCOMES:
Change in onset and sexual risk behaviors from baseline to 6 months | Up to 6-months
  Measures will ask youth to report a history of sexual intercourse and the age of onset, proportion of unprotected acts in past 30 days, frequency of condom use in past 30 days, condom use during the last episode, and number of sexual partners in past 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ismayilova, PhD, Principal Investigator — University of Chicago School of Social Service Administration
Locations (1):
- Columbia University Global Heath Research Center of Central Asia, Almaty, Kazakhstan

REFERENCES:
- [Result] Ismayilova L, Terlikbayeva A. Building Competencies to Prevent Youth Substance Use in Kazakhstan: Mixed Methods Findings From a Pilot Family-Focused Multimedia Trial. J Adolesc Health. 2018 Sep;63(3):301-312. doi: 10.1016/j.jadohealth.2018.04.005. Epub 2018 Jul 10. PMID 30006027
- [Result] Ismayilova L, Terlikbayeva A, Rozental Y. Computerized intervention to prevent drug use among at-risk adolescents in Central Asia: Preliminary family-level findings from a pilot mixed methods trial. Int J Drug Policy. 2019 Jun;68:75-85. doi: 10.1016/j.drugpo.2019.03.022. Epub 2019 Apr 16. PMID 31003194